CLINICAL TRIAL: NCT01687010
Title: Diagnostic and Prognostic Value of Combination Biomarkers in the Critically Ill Patient With Sepsis.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jianfeng Xie (Other)
Collaborators: Southeast University, China (Other)
Responsible Party: Sponsor-Investigator, Jianfeng Xie, Physician of critical care department, Southeast University, China
Organization: Southeast University, China (Other)
Other Study IDs: PCT001
Record Dates: First submitted 2012-09-13; First posted 2012-09-18 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2012-08

CONDITIONS: Diagnostic and Predictive Value
Keywords: CRP, PCT, IL-6, Diagnosis, Prediction
MeSH Terms: conditions — Disease

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Sepsis is a common cause for morbidity and mortality in critically ill patients. With the development of medical skills, the mortality is still remain very high. Inappropriateness of initial antibiotic treatment is an important risk factor for mortality and effective antimicrobial administration within the first hour of documented hypotension was associated with increased survival to hospital discharge in adult patients with septic shock. However, the early treatment based on early diagnosis.But it is very difficult to diagnosis because of lack of specific clinic symptom and sign.When severe sepsis occur, biomarker could be helpful to diagnosis. Unfortunately, the diagnostic value of single biomarker is limited. Therefore, combine several biomarkers could enhance the diagnostic value.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients admitted into ICU

Exclusion Criteria:

* Age younger than 18 years
* Refuse to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2012-03; Study Completion 2012-10 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Critical Care Medicine Nanjing Zhong-da Hospital Southeast University School of Medicine, Nanjing, Jiangsu, China